CLINICAL TRIAL: NCT06038994
Title: Prognostic Value of Surem TRAF3IP2 Level in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jin Geng, associate doctor, Nanjing Medical University
Other Study IDs: 20230901
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Myocardial Infarction, Acute
Keywords: TRAF3IP2, Myocardial Infarction, Coronary angiography, MACEs
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The blood sample will be collected, and the surem TRAF3IP2 levels will be measured using ELASA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute myocardial infarction who experienced CAG: Patients with acute myocardial infarction who experienced coronary angiography
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an obvertional study, and there is no intervention.

SUMMARY:
To evaluate the prognostic value of surem TRAF3IP2 levels in patients with acute myocardial infarction

DETAILED DESCRIPTION:
Previous study had concluded that TRAF3IP2 plays a causal role in atherosclerotic plaque development and vulnerability in mice. However, no human data was available. In the present study, patients diagnosed with acute myocardial infarction who receive coronary angiography will be enrolled. Their surem TRAF3IP2 levels will be tested using ELASA. The association of surem TRAF3IP2 levels with the major adverse cardiac events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute myocardial infarction
2. patients received coronary angiography
3. invasive management within 72 h of hospital admission

Exclusion Criteria:

1. NYHA III-IV
2. malignant tumor
3. acute infection
4. thyroid dysfunction
5. Life expectancy of b1 y
6. Unsuitable for PCI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute myocardial infarction who received coronary angiography well enrolled in Huai'an First People's Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
MACEs (major adverse cardiac events) | 1 year
  MACEs were defined as a composite of cardiac death, hospitalization for myocardial infarction or heart failure

SECONDARY OUTCOMES:
cardiac death | 1 year
  and death due to cardiac reasons, such as myocardial infarction or heart failure
hospitalization for myocardial infarction or heart failure | 1 year
  hospitalization for myocardial infarction or heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Shuren Ma, MD., Principal Investigator — NJMU
Locations (1):
- Huai'an First People's Hospital, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.